CLINICAL TRIAL: NCT05973669
Title: MED-EL Remote Care Multi-Center Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: US2302 MED-EL Remote Care
Record Dates: First submitted 2023-07-14; First posted 2023-08-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss, Sensorineural; Cochlear Implant; Cochlear Implant Recipients; Hearing Disorders; Cochlear Implants
Keywords: cochlear implants; telehealth; remote care
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Remote cochlear implant support (Experimental): Participants will use MED-EL Remote Care to test their hearing and device functionality. Participants and clinicians will complete user feedback surveys regarding their experience and time/cost-savings.
  Interventions: Device: MED-EL Remote Care

INTERVENTIONS:
Device: MED-EL Remote Care — Remote cochlear implant support

SUMMARY:
MED-EL Remote Care is a way for MED-EL cochlear implant users to check their hearing and cochlear implant device from any location, without the need for a scheduled, in-person appointment with their audiologist. This study will assess the effectiveness, efficiencies, and useability of MED-EL Remote Care.

DETAILED DESCRIPTION:
This prospective multicenter study will include MED-EL cochlear implant users from the US and Canada. This study will assess the effectiveness, efficiencies, and useability of MED-EL Remote Care.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with at least one MED-EL cochlear implant
* ≥ 2 weeks since activation of the cochlear implant
* Availability of existing aided Pediatric/AZ Bio (quiet and/or noise) and CNC word scores, or the ability to complete these at baseline
* Utilizing a compatible audio processor in the SONNET or RONDO product lines
* Ability to complete app-based hearing assessments
* Commitment to comply with all study procedures for the duration of the study
* Access to the internet via a smartphone that meets the following requirements:
* Android or iOS operating systems
* A smartphone supporting Bluetooth® 4.2 or higher
* A minimum of 200 MB free storage space

Exclusion Criteria:

* Inability or unwillingness to perform the requirements of the clinical investigation
* Unrealistic expectations regarding the possible benefits, risks, and limitations of remote cochlear implant care
* Inability of the subject or caregiver to demonstrate basic skills for operating a smartphone, computer, or app-based tasks after training by the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Remote Care Completion | Up to 6 months post-training
  Number and proportion of fully completed Remote Care visits.

SECONDARY OUTCOMES:
Patient time savings | Up to 6 months post-training
  Average time estimates associated with attending an in-clinic appointment compared to Remote Care completion time.
Patient cost estimates | Up to 6 months post-training
  Descriptive summaries of patient-estimated costs associated with attending an in-clinic appointment.
Clinician time savings | Up to 6 months post-training
  Average clinician-reported time estimates associated with in-clinic appointments compared to Remote Care completion time.
Patient Feedback Survey | Up to 6 months post-training
  Subject satisfaction measured using a custom questionnaire administered after each use of Remote Care. Each item is scored using a 5-point Likert scale with 1 always indicating a negative response and 5 a positive response. A total higher score indicates higher satisfaction.
Clinician Feedback Survey | Mid-enrollment to enrollment completion
  Clinician satisfaction measured using a custom questionnaire administered at mid-enrollment and at study completion. Each item is scored using a 5-point Likert scale with 1 always indicating a negative response and 5 a positive response. A total higher score indicates higher satisfaction.
Remote hearing assessments | Up to 6 months post-training
  Average remote hearing assessment results compared to standard aided test results obtained at baseline.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maruthurkkara S, Case S, Rottier R. Evaluation of Remote Check: A Clinical Tool for Asynchronous Monitoring and Triage of Cochlear Implant Recipients. Ear Hear. 2022 Mar/Apr;43(2):495-506. doi: 10.1097/AUD.0000000000001106. PMID 34320523
- [Background] Takano K, Kaizaki A, Kimura A, Nomura K, Yamazaki N, Shintani T, Himi T. Telefitting of Nucleus Cochlear Implants: A Feasibility Study. Am J Audiol. 2021 Mar 10;30(1):16-21. doi: 10.1044/2020_AJA-20-00041. Epub 2021 Feb 8. PMID 33555935
- [Background] Slager HK, Jensen J, Kozlowski K, Teagle H, Park LR, Biever A, Mears M. Remote Programming of Cochlear Implants. Otol Neurotol. 2019 Mar;40(3):e260-e266. doi: 10.1097/MAO.0000000000002119. PMID 30741905
- [Background] Cullington H, Kitterick P, Weal M, Margol-Gromada M. Feasibility of personalised remote long-term follow-up of people with cochlear implants: a randomised controlled trial. BMJ Open. 2018 Apr 20;8(4):e019640. doi: 10.1136/bmjopen-2017-019640. PMID 29678970
- [Background] Schepers K, Steinhoff HJ, Ebenhoch H, Bock K, Bauer K, Rupprecht L, Moltner A, Morettini S, Hagen R. Remote programming of cochlear implants in users of all ages. Acta Otolaryngol. 2019 Mar;139(3):251-257. doi: 10.1080/00016489.2018.1554264. PMID 31056039
- [Background] Hughes ML, Sevier JD, Choi S. Techniques for Remotely Programming Children With Cochlear Implants Using Pediatric Audiological Methods via Telepractice. Am J Audiol. 2018 Nov 19;27(3S):385-390. doi: 10.1044/2018_AJA-IMIA3-18-0002. PMID 30452743
- [Background] Eikelboom RH, Jayakody DM, Swanepoel DW, Chang S, Atlas MD. Validation of remote mapping of cochlear implants. J Telemed Telecare. 2014 Jun;20(4):171-177. doi: 10.1177/1357633X14529234. Epub 2014 Mar 27. PMID 24675003
- [Background] McElveen JT Jr, Blackburn EL, Green JD Jr, McLear PW, Thimsen DJ, Wilson BS. Remote programming of cochlear implants: a telecommunications model. Otol Neurotol. 2010 Sep;31(7):1035-40. doi: 10.1097/MAO.0b013e3181d35d87. PMID 20147864
- [Background] Ramos A, Rodriguez C, Martinez-Beneyto P, Perez D, Gault A, Falcon JC, Boyle P. Use of telemedicine in the remote programming of cochlear implants. Acta Otolaryngol. 2009 May;129(5):533-40. doi: 10.1080/00016480802294369. PMID 18649152